CLINICAL TRIAL: NCT05535335
Title: Brief-Illness Perception Questionnaire (Brief-IPQ) Used as Prediction of Outcome in Patients With Chronic Non-malignant Pain After Treatment in a Multidisciplinary Pain Clinic
Brief Title: Brief-Illness Perception Questionnaire (Brief-IPQ) Used in Patients With Chronic Non-malignant Pain
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: REG-1303-2022
Record Dates: First submitted 2022-03-24; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-03

CONDITIONS: Non-malignant Pain; Chronic Pain
Keywords: Placebo, chronic pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators wish to investigate if there are any difference in the BIPQ score in persons with chronic low back pain from admission to the Pain Centre at Zealand University Hospital Koege (ZUH), and when discharged.

DETAILED DESCRIPTION:
Chronic pain conditions are frequent in the danish population. More than 1.2 million Danes over the age of 16 are living with chronic pain. Chronic pain affects the health-related quality of life and functioning and is associated with reduced work ability, lost earnings and disability. At the Interdisciplinary Pain Center Zealand University Hospital Koege, Denmark, patients with chronic pain are received and treated based on the Bio-Psycho-Social Pain Model. The treatment of patients with complex chronic non-malignant pain can be complicated by psychological and / or social factors. The need for a screening of psychological factors in connection with the examination and planning of the pain management in the Interdisciplinary Pain Center is obvious as the patient's perception of illness and expectation of treatment have been shown to play a role in the treatment response. The Brief Illness Perception Questionnaire (Brief-IPQ) provides a quick assessment of the patient's disease perception and expectation of treatment and has proved useful in clinical practice. In this study, a Danish version of Brief-IPQ is used, which initially was taken from https://www.uib.no. Items as stated in research by L. van Oort et al (2011) have been adapted to the Danish version. A copy of the latest version can be obtained from Interdisciplinary Pain Center Zealand University Hospital Koege, Denmark.

The study:

Participants:

Patients with chronic low back pain admitted to the Pain Centre after June 2021 at ZUHK.

* Persons ≥18 years
* Persons who suffers from chronic back pain and are admitted to the Pain Centre at Zealand University Hospital in Køge, Denmark
* Persons who have completed the BIPQ both at first and at last visit in the Pain Centre

Numbers 100 patients with both pre and post admission IBPQ score

Timeframe The data will be analyzed when there is a full dataset on 100 patients admitted from June 2020

Location of the study The Pain Centre at Zealand University Hospital, Koege

The patients will answer the questionnaire including the following data online before visiting the pain Centre and after treatment. Thereby the investigators can estimate the result of treatment compared to the BIPQ score before entry to treatment statistically. and thereby generate estimates concerning the success of pain treatment measured by BIPQ.

* The Pain Self-Efficacy Questionnaire (PSEQ) is a 10-item questionnaire, to assess the confidence people with ongoing pain have in performing activities while in pain.
* Pain during movement is measured by the Numeric Rating Scale (NRS) from 0 to 10
* For measuring the patients fear of movement related pain (fear avoidance) the 17 items questionnaire Tampa Scale of Kinesiophobia (TSK) will be used.

  0= No pain at all and 10= worse imaginable pain
* Pain catastrophizing is measured by the Pain Catastrophizing Scale (PCS) and includes the following items rumination ("I can't stop thinking about how much it hurts"), magnification ("I worry that something serious may happen"), and helplessness ("There is nothing I can do to reduce the intensity of the pain"). The PCS total score is computed by summing responses to all 13 items. PCS total scores range from 0 - 52.
* Placebo measured with BIPQ. The BIPQ investigates the following; cognitive meaning (consequences, time perspective, personally control, treatment control and identity), emotional meaning (concerns, emotions), understanding of the condition and finally the patient´s own evaluation of the three most important reasons for the condition 8.

A decrease in BIPQ score will be defined as the mean +/- 1SD as cut-off.

All data will be derived from the PainData database. An examination is made of whether the patient meets the inclusion or exclusion criteria

• Data will be stored in an Excel file and the statistical analyses will performed using SPSS

Ethical aspects:

All information will be treated confidentially and all data will be anonymized by a secretary. The Investigator will keep an identification list of all patients who have been included. This list will include the patient's full name and CPR number. Collected data will be recorded in a Case Report Form. The results will be stored and analyzed using a computer and the anonymity of the patients will be preserved and local data law will be observed. Data will be stored in accordance with existing regulations. Data is stored in anonymized form and correlation and regression analysis will be performed after 6 months. The study is conducted in accordance with applicable clinical trial rules. Investigators are responsible for the handling and archiving of data in accordance with applicable rules in addition to the Act on the Processing of Personal Data and the Health Act. Data belong to the investigators. The project has been reported to the local ethic committee.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the multidisciplinary pain clinic at Zealand University Hospital with low back pain
* Understand Danish spoken and written

Exclusion Criteria:

* Patients with insufficient cognitive abilities
* Patients who decline to participate in the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with chronic non-malignant pain conditions reffered to the multidisciplinary pain clinic with low back pain
Sampling Method: Non-Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2020-06-06 (Actual); Primary Completion 2022-04-03 (Actual); Study Completion 2022-04-03 (Actual)

PRIMARY OUTCOMES:
Differences in illness perception | Change in Illness peception score Measured at admission and at discharge between the 12-6-2020 - 03-04-2022
  Change in Brief Illness perception will be measured by using the Brief Illness perception questionnaire. The IPQ-B consists of nine items rated on a scale from 0 (minimum) to 10 (maximum). Illness perception Scores 0-24, low scores, 24-56 moderate, 56- 80 high scores.

OTHER OUTCOMES:
Differences in Fear Avoidance | Change in Fear avoidance will be measured at admission and at discharge between the 12-6-2020 - 03-04-2022
  Change in Fear avoidance will be measured by using the 17 items Tampa Scale of Kinesiophobia, Scores range from 17 to 68. Low scores indicate no kinesiophobia and high scores extreme fear of pain with movement. Cut off score = 37.
Differences in Quality of life | Change in Quality of life will be measured at admission and at discharge between the 12-6-2020 - 03-04-2022
  Change in Quality of life will be measured by using the PROMIS-10 questionnaire.Using T-scores, median = 50, higher scores over 50 indicates wellbeeing.
Differences in Pain Self efficacy | Change in Pain Selv Efficacy will be measured at admission and at discharge between the 12-6-2020 - 03-04-2022
  Change in Pain Self efficacy will be measured by using the 2 items fra 10 item questionnaire: PSEQ. PSEQ 1 and PSEQ 2. numbers are calculated by summing the numbers. Median = 3, Scores higher than 3 means high confidence, lower than 3 means low confidence.
Differences in Pain Catastrophizing | Change in Pain Catastrophizing will be measured at admission and at discharge between the 12-6-2020 - 03-04-2022
  Change in Pain Catastrophizing will be measured by using the 13 items Pain Catastrophizing Scale. PCS range from 0 to 52. Subclinical = 0 to 29; Mild = 30 to 39; Moderate = 40 to 49; Severe = 50 to 59; Extreme = 60 to 100.
Differences in Numeric rating scale | Change in Pain intensity during movement measured at admission and at discharge between the 12-6-2020 - 03-04-2022
  Change in Pain intensity during movement measured from 0-10, where 10 is the worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Anja Geisler, phd., Study Director — Koge Universitets Hospital
Locations (1):
- Zealand University Hospital, Køge, Region Sjælland, Denmark